CLINICAL TRIAL: NCT04676412
Title: A Phase 3, Randomized, Double-blind Trial of Pembrolizumab (MK-3475) With or Without Lenvatinib (E7080/MK-7902) in Participants With Treatment-naïve, Metastatic Nonsmall Cell Lung Cancer (NSCLC) Whose Tumors Have a Tumor Proportion Score (TPS) Greater Than or Equal to 1% (LEAP-007)
Brief Title: Efficacy and Safety Study of Pembrolizumab (MK-3475) With or Without Lenvatinib (MK-7902/E7080) in Adults With Programmed Cell Death-Ligand 1 (PD-L1)-Positive Treatment-naïve Nonsmall Cell Lung Cancer (NSCLC) [MK-7902-007/E7080-G000-314/LEAP-007] - China Extension Study
Acronym: LEAP-007
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7902-007 China Extension; MK-7902-007 (Other: MSD); E7080-G000-314 (Other: Eisai Protocol Number); LEAP-007 (Other: MSD)
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Results first posted 2022-11-09 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death-ligand 1 (PD-L1, PDL1); programmed cell death-ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pembrolizumab + Lenvatinib (Experimental): Participants receive pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily (QD) on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib
- Pembrolizumab + Placebo (Active Comparator): Participants receive pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule QD on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Placebo for lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Lenvatinib — oral capsule
  Other Names: MK-7902; E7080; LENVIMA®
  Arms: Pembrolizumab + Lenvatinib
Drug: Placebo for lenvatinib — oral capsule
  Arms: Pembrolizumab + Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of pembrolizumab (MK-3475) combined with lenvatinib (MK-7902/E7080) compared to pembrolizumab alone (with placebo for lenvatinib) in treatment-naïve adults with no prior systemic therapy for their metastatic non-small cell lung cancer (NSCLC) whose tumors have a programmed cell death-ligand 1 (PD-L1) Tumor Proportion Score (TPS) greater than or equal to 1%.

The primary study hypotheses are that: 1) the combination of pembrolizumab and lenvatinib is superior to pembrolizumab alone as assessed by Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1); and 2) the combination of pembrolizumab and lenvatinib is superior to pembrolizumab alone as assessed by Overall Survival (OS).

DETAILED DESCRIPTION:
The main study will have a duration of approximately 5 years and the extension period will have a duration of approximately 1 year. The base study and the China extension to MK-7902-007 (NCT03829332) will enroll a total of approximately 120 Chinese participants.

As of 30-Jul-2021, active participants, investigator, and sponsor personnel or delegate(s) involved in the treatment administration or clinical evaluation of the participants will be unblinded. Participants will discontinue lenvatinib and placebo, and participants who remain on treatment will receive open-label pembrolizumab only.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC)
* Has Stage IV NSCLC (American Joint Committee on Cancer [AJCC])
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)
* Has tumor tissue that demonstrates programmed cell death-ligand 1 (PD-L1) expression in ≥1% of tumor cells (Tumor Proportion Score [TPS] ≥1%) as assessed by immunohistochemistry (IHC) 22C3 pharmDx assay (Dako North America, Inc.) at a central laboratory
* Has a life expectancy of ≥3 months
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days before the first dose of study treatment but before randomization
* Male participants must agree to the following during the treatment period and for ≥7 days after the last dose of lenvatinib/matching placebo: 1) Be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent, OR 2) Must agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause)
* Female participants are eligible to participate if not pregnant or breastfeeding, and ≥1 of the following applies: 1) Is not a woman of child-bearing potential (WOCBP), OR 2) Is a WOCBP and is using a highly effective contraceptive method that has a low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle during the treatment period and for ≥120 days post pembrolizumab or ≥30 days post lenvatinib/matching placebo, whichever occurs last
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mm Hg and no change in antihypertensive medications within 1 week before randomization
* Has adequate organ function

Exclusion Criteria:

* Has known untreated central nervous system metastases and/or carcinomatous meningitis
* Has a known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for ≥3 years since initiation of that therapy (Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.)
* Has radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation
* Has an active autoimmune disease that has required systemic treatment in the past 2 years Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Has had an allogeneic tissue/solid organ transplant
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a history of (noninfectious) pneumonitis that required systemic steroids or current pneumonitis/interstitial lung disease
* Has a known history of hepatitis B or known active hepatitis C virus infection
* Has a history of a gastrointestinal condition or procedure that in the opinion of the investigator may affect oral study drug absorption
* Has significant cardiovascular impairment within 12 months of the first dose of study treatment, such as a history of congestive heart failure greater than New York Heart Association Class II, unstable angina, myocardial infarction, cerebrovascular accident/stroke, or cardiac arrhythmia associated with hemodynamic instability
* Has not recovered adequately from any toxicity and/or complications from major surgery before starting study treatment
* Has a known history of active tuberculosis (TB)
* Has an active infection requiring systemic therapy
* Has previously had a severe hypersensitivity reaction to treatment with a monoclonal antibody or has a known sensitivity or intolerance to any component of lenvatinib or pembrolizumab
* Has received prior systemic chemotherapy or other targeted or biological antineoplastic therapy for their metastatic NSCLC
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], Tumor necrosis factor receptor superfamily, member 4 [OX 40], tumor necrosis factor receptor superfamily member 9 [CD137]) or has received lenvatinib as monotherapy or in combination with anti- programmed cell death protein (anti-PD-1) agents
* Has received radiotherapy within 14 days before the first dose of study treatment or received lung radiation therapy of >30 Gray (Gy) within 6 months before the first dose of study treatment. (Note: Participants must have recovered from all radiation-related toxicities to ≤Grade 1, not require corticosteroids, and not have had radiation pneumonitis.)
* Has a diagnosis of immunodeficiency or is receiving any form of immunosuppressive therapy within 7 days before the first dose of study treatment
* Is receiving systemic steroid therapy (doses >10 mg daily of prednisone equivalent) within 7 days before the first dose of study treatment
* Has received a live vaccine within 30 days before the first dose of study treatment
* Has had major surgery within 3 weeks prior to first dose of study treatment
* Has pre-existing ≥Grade 3 gastrointestinal or non-gastrointestinal fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (17):
- China (17):
  - Anhui Provincial Hospital ( Site 0108), Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University ( Site 0113), Hefei, Anhui
  - Peking Union Medical College Hospital ( Site 0105), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0102), Beijing, Beijing Municipality
  - Beijing Chest Hospital Capital Medical University ( Site 0111), Beijing, Beijing Municipality
  - Xiangya Hospital of Central South University ( Site 0115), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 0104), Changsha, Hunan
  - Zhongshan Hospital Fudan University ( Site 0100), Shanghai, Hunan
  - Jiangsu Cancer Hospital ( Site 0101), Nanjing, Jiangsu
  - The First Hospital of Jilin University ( Site 0110), Changchun, Jilin
  - Shanghai Chest Hospital ( Site 0112), Shanghai, Shanghai Municipality
  - 1st Affil Hosp of Med College of Xi'an Jiaotong University ( Site 0103), XiAn, Shanxi
  - West China Hospital of Sichuan University ( Site 0117), Chengdu, Sichuan
  - The First Affiliated Hospital Zhejiang University ( Site 0106), Hangzhou, Zhejiang
  - Hangzhou First People's Hospital ( Site 0109), Hangzhou, Zhejiang
  - 2nd Affil Hosp of Zhejiang University College of Medicine ( Site 0114), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0116), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Yang JC, Han B, De La Mora Jimenez E, Lee JS, Koralewski P, Karadurmus N, Sugawara S, Livi L, Basappa NS, Quantin X, Dudnik J, Ortiz DM, Mekhail T, Okpara CE, Dutcus C, Zimmer Z, Samkari A, Bhagwati N, Csoszi T. Pembrolizumab With or Without Lenvatinib for First-Line Metastatic NSCLC With Programmed Cell Death-Ligand 1 Tumor Proportion Score of at least 1% (LEAP-007): A Randomized, Double-Blind, Phase 3 Trial. J Thorac Oncol. 2024 Jun;19(6):941-953. doi: 10.1016/j.jtho.2023.12.023. Epub 2023 Dec 29. PMID 38159809
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 107 Chinese participants were randomized and received treatment (global study [NCT03829332; n=80] or to the extension portion [n=27]).
Groups:
- Pembrolizumab + Lenvatinib: Participants received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily (QD) on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity. As of 30-Jul-2021, participants discontinued lenvatinib and participants who remained on treatment received open-label pembrolizumab only at same dose and schedule.
- Pembrolizumab + Placebo: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule QD on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity. As of 30-Jul-2021, participants discontinued placebo and participants who remained on treatment received open-label pembrolizumab only at same dose and schedule.
Period: Overall Study
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Started | 49 | 58
Completed | 0 | 0
Not Completed | 49 | 58
Not completed — Death | 28 | 31
Not completed — Lost to Follow-up | 1 | 2
Not completed — Sponsor Decision | 20 | 23
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: All Chinese participants who were randomized to the global study (NCT03829332) or to the extension portion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo | Total
Number analyzed (Participants) | 49 | 58 | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (8.2) | 64.2 (7.6) | 64.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 42 | 48 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 58 | 107
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 49 | 58 | 107
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
  Participants
    ECOG=0 | 6 | 10 | 16
    ECOG=1 | 43 | 48 | 91
Programmed Cell Death Ligand 1 (PD-L1) Status at Baseline [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Randomization of participants in the study was stratified by PD-L1 tumor proportion score (TPS) at baseline (1-49% or ≥ 50%). Higher percentages of PD-L1 TPS staining correspond to higher positivity of PD-L1 on a tumor.
  Participants
    TPS=1-49% | 21 | 33 | 54
    TPS≥ 50% | 28 | 25 | 53
Geographic Region [Count of Participants; unit: Participants] — Randomization of participants in this study was stratified by geographic region of the enrolling site (East Asia or non-East Asia).
  Participants
    East Asia | 49 | 58 | 107
    Non-East Asia | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR
Description: ORR was defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experienced CR or PR as assessed by BICR were presented.
Time Frame: Up to approximately 18 months
Population: All Chinese participants who were randomized to the global study (NCT03829332) or to the extension portion that were evaluable for response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 42 | 53
Percentage of participants | 33.3 [19.6 to 49.5] | 39.6 [26.5 to 54.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — Percent difference and 95% CI were calculated using Miettinen and Nurminen method with Efron's method of tie handling with treatment as a covariate stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and baseline PD-L1 status (1-49% versus ≥50%); p = 0.79262, Stratified Miettinen and Nurminen; One-sided p-value for testing. H0: difference in percentage =0 versus H1: difference in percentage > 0; Difference in percentage = -8.4, 95% CI 2-sided [-27.4 to 11.9]

2. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced an AE were reported.
Time Frame: Up to approximately 52 months
Population: All Chinese participants who were randomized to the global study (NCT03829332) or to the extension portion who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 58
Participants | 49 | 57

3. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinued study treatment due to an AE were reported
Time Frame: Up to approximately 30 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 58
Participants | 19 | 13

4. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Combined Global Health Status / Quality of Life (Items 29 & 30) Scale Combined Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall quality of life (QoL) of cancer patients. Participant responses to questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and QoL ("How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) is computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. Per protocol, the change from baseline in GHS and QoL combined score was presented.
Time Frame: Baseline and Week 21
Population: All Chinese participants who were randomized to the global study (NCT03829332) or to the extension portion who received at least one dose of treatment and had at least one EORTC-QLQ-C30 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Score on a scale | -2.43 [-8.69 to 3.83] | -2.18 [-8.34 to 3.98]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — Difference in LS means and 95% CI were calculated using the Constrained longitudinal data analysis (cLDA) model with covariates for treatment by study visit interaction & stratified by ECOG performance status (0 versus 1) and baseline PD-L1 Status (1% to 49% versus >=50%); p = 0.9519, cLDA model; Two-sided p-value based on cLDA model with covariates for treatment by study visit interaction; stratified by ECOG and baseline PDL-1; Difference in Least Square (LS) Means = -0.25, 95% CI 2-sided [-8.59 to 8.09]

5. Secondary Outcome: Change From Baseline in Cough (EORTC Quality of Life Questionnaire-Lung Cancer Module 13 [QLQ-LC13] Item 31) Score
Description: The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in cough (EORTC QLQ-LC13 Item 31) score will be presented. A lower score indicates a better outcome.
Time Frame: Baseline and Week 21
Population: All Chinese participants who were randomized to the global study (NCT03829332) or to the extension portion who received at least one dose of treatment and had at least one assessment for EORTC QLQ-LC13 available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Score on a scale | -2.97 [-9.97 to 4.04] | -11.78 [-18.64 to -4.92]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — Difference in LS means and 95% CI were calculated using the cLDA model with covariates for treatment by study visit interaction & stratified by ECOG performance status (0 versus 1) and baseline PD-L1 Status (1% to 49% versus >=50%); p = 0.0628, cLDA model; [statistical method as in outcome 4, analysis 1]; Difference in LS Means = 8.81, 95% CI 2-sided [-0.49 to 18.11]

6. Secondary Outcome: Change From Baseline in Chest Pain (EORTC QLQ-LC13 Item 40) Score
Description: The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in chest pain (EORTC QLQ-LC13 Item 40) score was reported. A lower score indicated a better outcome.
Time Frame: Baseline and Week 21
Population: All Chinese participants who were randomized to the global study (NCT03829332) or to the extension portion who received at least one dose of treatment and had at least one EORTC QLQ-LC13 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Score on a scale | -3.84 [-9.95 to 2.28] | -7.42 [-13.41 to -1.44]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.3298, cLDA model; [statistical method as in outcome 4, analysis 1]; Difference in LS Means = 3.59, 95% CI 2-sided [-3.70 to 10.87]

7. Secondary Outcome: Change From Baseline in Dyspnea (EORTC QLQ-C30 Item 8) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in dyspnea (EORTC QLQ-C30 Item 8) score was reported. A lower score indicated a better outcome.
Time Frame: Baseline and Week 21
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Score on a scale | 0.54 [-7.85 to 8.94] | 0.82 [-7.41 to 9.06]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.9594, cLDA model; [statistical method as in outcome 4, analysis 1]; Difference in LS Means = -0.28, 95% CI 2-sided [-11.32 to 10.75]

8. Secondary Outcome: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. Per protocol, the change from baseline in EORTC QLQ-C30 physical functioning (Items 1-5) combined score was presented.
Time Frame: Baseline and Week 21
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Score on a scale | -5.15 [-10.78 to 0.48] | 0.38 [-5.08 to 5.84]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.1620, cLDA model; [statistical method as in outcome 4, analysis 1]; Difference in LS Means = -5.53, 95% CI 2-sided [-13.37 to 2.31]

9. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-C30 Combined Global Health Status /Quality of Life (Items 29 & 30) Scale Combined Score
Description: EORTC QLQ-C30 is a questionnaire to assess QoL of cancer patients. Participant responses to questions on GHS ("How would you rate your overall health during the past week?") and QoL ("How would you rate your overall QoL during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) was computed by averaging raw scores of the 2 items and applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in GHS-QoL combined score. A longer TTD indicates a better outcome.
Time Frame: Up to approximately 25 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Months | NA [5.7 to NA] — NA = Median and upper limit was not reached due to insufficient number of participants with an event. | NA [8.9 to NA] — NA = Median and upper limit was not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — HR and 95% CI were based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG performance status (0 versus 1) and baseline PD-L1 status (1-49% versus ≥50%); p = 0.9419, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG performance status and baseline PD-L1 status; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.47 to 2.26]

10. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-LC13 Cough (Item 31) Scale Score
Description: EORTC QLQ-LC13 is a lung cancer specific questionnaire. Participant responses to the question: "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0-100. A lower score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in cough (Item 31). A longer TTD indicates a better outcome.
Time Frame: Up to approximately 25 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Months | NA [NA to NA] — NA = Median, lower limit, and upper limit were not reached due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, lower limit, and upper limit were not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — HR and 95% CI were calculated using Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG performance status (0 versus 1) and baseline PD-L1 status (1-49% versus ≥50%); p = 0.9789, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG performance status and baseline PD-L1 status; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.43 to 2.38]

11. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-LC13 Chest Pain (Item 40) Scale Score
Description: EORTC QLQ-LC13 is a lung cancer specific questionnaire. Participant responses to the question: "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0-100. A lower score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in cough (Item 40). A longer TTD indicates a better outcome.
Time Frame: Up to approximately 25 months
Population: All Chinese participants who were randomized to the global study (NCT03829332) or to the extension portion who received at least one dose of treatment and had at least one EORTC-QLQ-LC13 assessment data available.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Months | NA [NA to NA] — NA = Median, lower limit, and upper limit were not reached due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, lower limit, and upper limit were not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.8856, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG performance status and baseline PD-L1 status; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.36 to 3.28]

12. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-C30 Dyspnea (Item 8) Scale Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to the question: "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in dyspnea (Item 8). A longer TTD indicates a better outcome.
Time Frame: Up to approximately 25 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Months | NA [5.8 to NA] — NA = Median and upper limit were not reached due to insufficient number of participants with an event. | NA [8.9 to NA] — NA = Median and upper limit were not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.3264, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG performance status and baseline PD-L1 status; Hazard Ratio (HR) = 1.55, 95% CI 2-sided [0.64 to 3.75]

13. Secondary Outcome: Time to True Deterioration (TTD) in the Composite Endpoint of EORTC QLQ-LC13 Cough (Item 31), EORTC QLQ-LC13 Chest Pain (Item 40), or EORTC QLQ-C30 Dyspnea (Item 8)
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients, including a single-item scale score for dyspnea (Item 8; score range:1=Not at All to 4=Very Much). Used in combination with QLQ-C30, the EORTC QLQ-LC13 is a supplemental lung cancer-specific module, including a single-item scale score for cough (Item 31; score range:1=Not at All to 4=Very Much ) and chest pain (Item 40, score range: 1=Not at All to 4=Very Much). The combined score of items 31, 40 and 8 was computed by averaging the raw scores of the items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. The TTD in the composite endpoint of EORTC QLQ-LC13 Item 31, EORTC QLQ-LC13 Item 40, EORTC QLQ-C30 Item 8 scale score was presented, defined as the time to first onset of a ≥10point decrease from baseline in anyone of the three scale items. A longer TTD indicates better outcome.
Time Frame: Up to approximately 25 months
Population: All Chinese participants who were randomized to the global study (NCT03829332) or to the extension portion who received at least one dose of treatment and had at least one EORTC-QLQ-C30 or EORTC QLQ-LC13 assessment data available.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Months | 5.78 [2.79 to NA] — NA = Upper limit was not reached due to insufficient number of participants with an event. | NA [3.45 to NA] — NA = Median and upper limit were not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.4068, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG performance status and baseline PD-L1 status; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.70 to 2.46]

14. Secondary Outcome: Time to True Deterioration (TTD) Based on Change From Baseline in EORTC QLQ-C30 Physical Functioning (Items 1-5) Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in physical functioning (Items 1 to 5). A longer TTD indicates a better outcome.
Time Frame: Up to approximately 25 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 49 | 55
Months | NA [6.2 to NA] — NA = Median and upper limit were not reached due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, lower limit, and upper limit were not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.0020, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG performance status and baseline PD-L1 status; Hazard Ratio (HR) = 7.81, 95% CI 2-sided [1.71 to 35.62]

15. Primary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from date of randomization to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. Data were from the product-limit (Kaplan-Meier) method for censored data. PFS as assessed by BICR per RECIST 1.1 was presented.
Time Frame: Up to approximately 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 42 | 53
Months | 6.1 [4.2 to 8.7] | 10.3 [5.6 to NA] — Upper limit of PFS not reached, due to insufficient number of participants with events in the study.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other — Hazard ratio (HR) and 95% confidence interval (CI) were calculated using Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and baseline PD-L1 status (1-49% versus ≥50%); p = 0.71084, Stratified Log Rank; One-sided p-value based on log-rank test stratified by ECOG performance status, geographic region of enrolling site and baseline PD-L1 status; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.61 to 2.25]

16. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to date of death from any cause.
Time Frame: Up to approximately 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 42 | 53
Months | 11.4 [8.4 to NA] — Upper limit of OS not reached, due to insufficient number of participants with death events in the study. | NA [NA to NA] — Median OS, Lower and Upper limit of OS not reached, due to insufficient number of participants with death events in the study.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; HR and 95% CIs were calculated using Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and baseline PD-L1 status (1-49% versus ≥50%); Test type: Other; p = 0.81970, Stratified Log Rank; [statistical method as in outcome 15, analysis 1]; Hazard Ratio (HR) = 1.53, 95% CI 2-sided [0.61 to 3.87]

ADVERSE EVENTS:
Time Frame: Up to approximately 52 months
Description: All-Cause Mortality includes all randomized participants. Serious and Other adverse events (AEs) includes all randomized participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Groups:
- Lenvatinib + Pembrolizumab: Participants received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily (QD) on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity. As of 30-Jul-2021, participants discontinued lenvatinib and participants who remained on treatment received open-label pembrolizumab only at same dose and schedule.
- Placebo + Pembrolizumab: Participants received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily (QD) on Days 1-21 of each 3-week cycle until progressive disease or unacceptable toxicity. As of 30-Jul-2021, participants discontinued placebo and participants who remained on treatment received open-label pembrolizumab only at same dose and schedule.
Arm/Group | Lenvatinib + Pembrolizumab | Placebo + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 28/49 | 32/58
Serious Adverse Events (participants affected / at risk) | 24/49 | 17/58
Other Adverse Events (participants affected / at risk) | 49/49 | 54/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=49) | Placebo + Pembrolizumab (N=58)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (3) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Coagulation time prolonged (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=49) | Placebo + Pembrolizumab (N=58)
Anaemia (Blood and lymphatic system disorders) | 14 (21) | 16 (31)
Arrhythmia (Cardiac disorders) | 4 (4) | 3 (4)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 8 (12)
Hypothyroidism (Endocrine disorders) | 22 (42) | 11 (12)
Abdominal distension (Gastrointestinal disorders) | 3 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 5 (5)
Constipation (Gastrointestinal disorders) | 3 (4) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 20 (38) | 8 (9)
Nausea (Gastrointestinal disorders) | 3 (4) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 5 (10) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (8) | 5 (8)
Asthenia (General disorders) | 4 (4) | 3 (3)
Chest discomfort (General disorders) | 3 (4) | 1 (1)
Chest pain (General disorders) | 6 (8) | 3 (3)
Fatigue (General disorders) | 5 (5) | 2 (2)
Malaise (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 10 (13) | 11 (14)
COVID-19 (Infections and infestations) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4)
Urinary tract infection (Infections and infestations) | 6 (16) | 8 (19)
Alanine aminotransferase increased (Investigations) | 14 (21) | 13 (21)
Amylase increased (Investigations) | 6 (12) | 3 (7)
Aspartate aminotransferase increased (Investigations) | 17 (27) | 16 (27)
Bilirubin conjugated increased (Investigations) | 4 (12) | 4 (5)
Blood alkaline phosphatase increased (Investigations) | 5 (6) | 1 (1)
Blood bilirubin increased (Investigations) | 9 (18) | 6 (12)
Blood creatinine increased (Investigations) | 6 (7) | 5 (6)
Blood glucose increased (Investigations) | 4 (6) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 4 (4)
Blood thyroid stimulating hormone increased (Investigations) | 12 (15) | 1 (2)
Blood urea increased (Investigations) | 6 (11) | 0 (0)
Blood urine present (Investigations) | 3 (7) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 5 (8) | 3 (5)
Lipase increased (Investigations) | 6 (12) | 2 (3)
Neutrophil count decreased (Investigations) | 4 (5) | 1 (1)
Platelet count decreased (Investigations) | 13 (19) | 4 (30)
Protein urine present (Investigations) | 3 (5) | 1 (4)
Urinary occult blood positive (Investigations) | 3 (3) | 3 (9)
Weight decreased (Investigations) | 21 (27) | 2 (3)
Weight increased (Investigations) | 3 (3) | 11 (17)
White blood cell count decreased (Investigations) | 6 (8) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 14 (19) | 8 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (14) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (6)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (8) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (12) | 8 (15)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7) | 7 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (8) | 6 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Hypoproteinaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (10) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (3)
Dizziness (Nervous system disorders) | 1 (2) | 4 (4)
Headache (Nervous system disorders) | 3 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3)
Haematuria (Renal and urinary disorders) | 10 (15) | 10 (16)
Proteinuria (Renal and urinary disorders) | 26 (48) | 11 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 7 (9)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 10 (26)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 (10) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (11) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 13 (21) | 7 (10)
Hypertension (Vascular disorders) | 21 (23) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT04676412/Prot_SAP_002.pdf